CLINICAL TRIAL: NCT05713435
Title: Use of Fractional CO2 Laser Versus Erbium:YAG Laser for the Treatment of Genitourinary Syndrome of Menopause (GSM) in Patients Using Aromatase Inhibitors: Double Blinded Randomized Controlled Clinical Trial.
Brief Title: Use of Fractional CO2 Laser Versus Erbium:YAG Laser for the Treatment of GSM in Patients Using Aromatase Inhibitors
Acronym: LASI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S66520
Record Dates: First submitted 2023-01-09; First posted 2023-02-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: genitourinary syndrome of menopause; intravaginal laser; breast cancer; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 3 parallel arms of equal size, participants can cross over after 3 initial treatments
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and outcome assessor are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mona Lisa Touch CO2 laser (Active Comparator): 1. Power: 30 W.
  2. Dwell time: 1000 μs.
  3. Spacing: 1000 μm.
  4. Depth: SmartStack parameter from 1 to 3 depending on the treatment status.
  5. D-pulse mode.
  6. At the introitus the power will be reduced to 24 W
  Interventions: Device: intravaginal laser
- Fotona Smooth erbium:YAG laser (Active Comparator): 1. Phase I (vaginal) Renovalase™ mode with (a) fluence of 5,5J/cm2, (b) SMOOTHTM mode frequency 1.6 Hz, and (c) spot size 7 mm.
  2. Phase II (vestibulum and introitus) Renovalase™ mode with (a) fluence 10 J/cm2, (b) SMOOTHTM mode frequency 1.6Hz, and (c) spot size 7 mm.
  Interventions: Device: intravaginal laser
- sham treatment (Sham Comparator): 1. The blocking device is inserted over the laser outlet before attaching the application speculum. With this device the laser beam is blocked entirely.
  2. Phase I (vaginal) Renovalase™ mode with (a) fluence of 5,5J/cm2, (b) SMOOTHTM mode frequency 1.6 Hz, and (c) spot size 7 mm.
  3. Phase II (vestibulum and introitus) Renovalase™ mode with (a) fluence 1,5 J/cm2, (b) SMOOTHTM mode frequency 1.6Hz, and (c) spot size 7 mm.
  Interventions: Device: intravaginal laser

INTERVENTIONS:
Device: intravaginal laser — application of intravaginal laser

SUMMARY:
To study the efficacy and safety of intravaginal CO2 laser versus intravaginal Er:YAG laser and sham application in alleviating genitourinary symptoms in patients receiving an aromatase inhibitor as adjuvant treatment of breast cancer

DETAILED DESCRIPTION:
The objective is to compare microablative fractional CO2 laser (CO2 laser) (SmartXide2 V2 LR, Monalisa Touch; DEKA, Florence, Italy) and non-ablative photothermal Erbium:YAG laser (Er:YAG laser) (Fotona Smooth™ XS; Fotona, Ljubljana, Slovenia) - with sham vaginal applications for treatment of vaginal dryness as the leading symptom in breast cancer patients with iatrogenic menopause and treated with an AI.

ELIGIBILITY:
Inclusion Criteria:

Recruited participants will meet all of these criteria:

* a history of breast cancer
* premenopausal at diagnosis of breast cancer
* using AI as an adjuvant treatment
* moderate to severe symptoms of GSM (VAS ≥ 4/10)
* currently menopausal, which can be either biochemical menopause as confirmed after chemotherapy, surgical or medicinally induced (GnRH analogues for the duration of the trial)

Exclusion Criteria:

* Not willing to abstain from vaginal intercourse for 1 week following laser therapy
* Use of non-hormonal vaginal preparations within the last 6 weeks before inclusion
* Use of hormonal therapy within 6 months prior to inclusion (systemic or local)
* Acute urinary or genital tract infections
* A history of genital fistula, a thin rectovaginal septum as determined by the investigator, or history of fourth degree laceration
* Prolapse ≥ grade 2 according to the Pelvic Organ Prolapse Quantification System
* Previous vaginal mesh implantation
* Abnormal result in the last cervical smear (maximum 36 month before enrollment)
* Active cancer treatment (radiotherapy or chemotherapy) ongoing or planned prior to the measurement of the primary outcome (6 months after inclusion, 3 months after last laser)
* Vaginal stenosis that does not allow the placement of the laser probe
* Any condition that could interfere with study compliance

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change in severity dryness as most bothersome symptom (MBS) of GSM at 3 months after the end of treatment | at 3 months after the end of treatment
  scored on a 10 cm VAS

SECONDARY OUTCOMES:
Patient reported effect of laser on other GSM symptoms | at 3 months after the end of treatment
  scored on a 10 cm VAS
Female Sexual Function Index (FSFI) | at 3 months after the end of treatment
  measured with FSFI questionnaire. The cut-off score of >26,55 will be used to discriminate between women with impaired and unimpaired sexual functioning
Urinary Distress Index (UDI-6) | at 3 months after the end of treatment
  Measured with UDI-6 questionnaire
The degree of discomfort of the treatment procedure by the participant | at the end of the each treatment-visit
  scored on a 10 cm VAS
The longevity of the effect | at 24 months after the end of treatment
  Determined by questioning the need the participant feels for repeat treatment, and its nature (repeat laser or alternatives) until two years after the end of treatment.
Vaginal pH | at 3 months after the end of treatment
  Measured with a pH indicator strip (range 3.6-6.1) and is sampled from the lateral vaginal wall in the lower third of the vagina
Vaginal Health Index Score (VHIS) | at 3 months after the end of treatment
  Scoring of vaginal moisture, vaginal fluid volume, vaginal elasticity, vaginal pH, and vaginal epithelial integrity on a scale of 1 (poorest) to 5 (best) according to the methods of Robert Wood Johnson Medical School. The lower the score, the greater the atrophy. Vaginal moisture is an assessment of the appearance and spread or consistency of the secretions which coat the vagina. Vaginal elasticity is a measure of the ability of the vaginal tissue to stretch from the examiner's finger. Vaginal epithelial integrity takes into account color, thickness, and ability of the tissue to resist breaking secondary to touch.
Vaginal Maturation Value (VMV) | at 3 months after the end of treatment
  A vaginal smear will be obtained from the lateral vaginal wall using a spatula and will be stained according to the Papanicolaou technique. The Vaginal Maturation Index (VMI) is evaluated by defining the proportion of superficial, intermediate, and parabasal epithelial cells on the smear. To combine this information into a single score for quantifying estrogenization, the VMV was calculated. It is based on weighted proportions of cell types from the VMI and calculated using Meisels' formula: the percentage of superficial cells (S) plus 0.5 times the percentage of intermediate cells (I) coded from the cytology sample [MV= %S + (0.5 × % I)
Description of adverse events | until 1 month after the last treatment visit
  Adverse events are questioned at each visit following an intravaginal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Housmans, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No